CLINICAL TRIAL: NCT03193775
Title: Impact of Hepatitis B Vaccination on HBsAg Kinetics, Interferon-inducible Protein 10 Level and Recurrence of Viremia
Brief Title: Impact of Hepatitis B Vaccination on HBs Antigenemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Amr Shaaban Hanafy, Assistant professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3777
Record Dates: First submitted 2017-05-26; First posted 2017-06-21 (Actual); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: HBV
Keywords: HBV vaccine; persistent; HBsAg; IP-10

STUDY DESIGN:
Intervention Model Description: Group I: inactive carriers (n=100). Group II: CHB exposed to nucleos(t)ides (n=120) till 6 months after HBe seroconversion and HBV DNA disappearance in HBeAg positive (n=60) or DNA disappearance in HBeAg negative patients (n=60). All showed persistent HBs antigenemia.
  -A control group (n=100) did not receive HBV vaccine
Masking Description: open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chronic HBV with persistent HBsAg (Active Comparator): inactive carriers (n=100). Group II: CHB exposed to nucleos(t)ides (n=120) till 6 months after HBe seroconversion and HBV DNA disappearance in HBeAg positive (n=60) or DNA disappearance in HBeAg negative patients (n=60). All showed persistent HBs antigenemia.
  they were given 30 µg of HBV vaccine initiated 6 months after HBe seroconversion and disappearance of HBV DNA.
  Interventions: Biological: HBV vaccine
- control group (No Intervention): A control group (n=100) did not receive HBV vaccine

INTERVENTIONS:
Biological: HBV vaccine — HBV vaccine which contains Purified HBsAg produced by recombinant DNA technology (Euvax-B, LG Life sciences, Korea) intramuscularly in deltoid region at three different time intervals (0, 1, 6 months).
  Arms: chronic HBV with persistent HBsAg

SUMMARY:
* HBV is not curable with persistent HBsAg even after the disappearance of HBV DNA.
* HBsAg > 1000 IU/ml is associated with the risk of virological recurrence and HCC.
* There is an impaired immune response to HBsAg and HBV vaccine is an easily available, cost-effective, non-harmful method of stimulating immunity.

DETAILED DESCRIPTION:
Persistent HBs antigenemia >1000 IU/ml has a possibility of viral reactivation and hepatoma in 8%; the effect of HBV vaccine on HBsAg was investigated, recurrence of viremia, insulin resistance, and fibrosis regression.

From August 2011 to October 2016, 220 participants with chronic hepatitis B were evaluated at the hepatology clinic-Internal medicine department-Zagazig university-Egypt. They were enrolled after approval of the ethical committee of Zagazig university hospital. Written informed consent was obtained for the interview, clinical evaluation, and blood sampling.

participants were divided into two groups:

* Inactive carriers (n=100) who were presented with persistent HBsAg, undetected HBV DNA, normal liver enzymes, positive HBeAb and had never been exposed to antiviral therapy.
* Patients exposed to NAs (n=120): tenofovir 300mg (n=65) or Entecavir 1mg (n=55): A- HBeAg-positive patients (n=60) who received NAs until 1 year after HBe seroconversion and disappearance of HBV DNA with persistent HBsAg B- HBeAg-negative patients (n=60) who received NAs till 3 years after the disappearance of HBV DNA; all showed persistent HBsAg.
* Exclusion criteria Clinically decompensated liver cirrhosis; hepatocellular carcinoma; other causes of liver disease or mixed causes (excessive alcohol consumption, autoimmune liver disease, immunosuppressive drugs, or who had been infected with hepatitis C virus.

B- Vaccination schedule

* All the participants had received 30 µg of recombinant HBV vaccine which contains Purified HBsAg produced by recombinant DNA technology (Euvax-B, LG Life Sciences, Korea) intramuscularly in the deltoid region at three different time intervals (0, 1, 6 months). The first dose of the vaccine was initiated 1 year after HBe seroconversion and disappearance of HBV DNA in HBe +ve or 3 years after the disappearance of HBV DNA in HBe -ve patients or immediately after diagnosis of inactive carriers. NAs were stopped three months after the 3rd dose of HBV vaccine
* Three months after the last dose of vaccine, the participants were evaluated for IP-10 level, the production of protective HBsAb, recurrence of viremia by regular HBV DNA, HBsAg quantification.

Patients who failed to produce HBsAb i.e. HBsAb titer < 10 IU/ml, were given a fourth booster dose of vaccination immediately after confirmation of vaccine non-response.

C- Control Group It included 100 participants who had CHB, with undetectable HBV DNA with persistence of HBsAg and they did not receive HBV vaccine. They were divided into treatment naïve (n=50) and treatment experienced (n=50) who were given tenofovir (n=30) or entecavir (n=20) which were stopped 3 years after HBV DNA disappearance and HBeAg seroconversion and followed for 3 years by evaluation of HBsAg level and HBV DNA every 6 months to detect the natural rate of HBV reactivation.

D- Laboratory analysis It included complete Blood Count, liver function tests, prothrombin time, prothrombin concentration (%), kidney function tests.

* HCV antibody, HBeAg, HBeAb, HBcAb.
* Real-time Quantitative PCR for HBV DNA was done at the baseline and then every 6 months after the last dose of HBV vaccine for 3 years (COBAS AMPLICOR HBV MONITOR, with a detection limit of 15 IU/ml; Roche Diagnostic Systems).
* Insulin resistance was done before initiation of vaccination and 3 months after the last dose of vaccination. It was calculated by HOMA-IR, a value greater than 2 indicates insulin resistance [20].
* HBV genotyping was performed using INNO-LiPA HBV Genotyping assay; Innogenetics NV, Ghent, Belgium.
* Determination of HBsAg titer (Elecsys HBsAg II assay, Roche Diagnostics, USA) [21]. It was done before vaccination and 3 months after the last dose of vaccine then every 6 months for 3 years.
* Anti-HBs antibodies were performed 3 months following the third dose of the vaccine or 3 months after the 4th booster dose. Seroconversion was considered if anti-HBs levels were above 10 IU/ml and non-response if anti-HBs levels were below 10 IU/ml [22].
* Serum IP-10 levels were determined in serum before vaccination and 3 months after the last dose of vaccine, by a solid-phase sandwich ELISA (Quantikine, R&D Systems, USA) (reference value: 7.8-500 pg/ml).

E- Abdominal ultrasonography participants were examined after 6 hours fast. Criteria of cirrhosis, portal hypertension, and the presence of fatty liver disease were documented.

F- Liver stiffness assessment (LSM) Fibroscan was performed to measure liver stiffness before antiviral therapy and 3 months after the last dose of HBV vaccine, with the number of shots is 10, interquartile range≤ 25%. Liver stiffness 2.5-7 kPa denotes (F0-1), 7-9.5 kPa (F2), 9.5-12.5 kPa (F3), >12.5 kPa denotes cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* HBV patients with persistent HBs antigenemia

Exclusion Criteria:

* decompensated liver cirrhosis
* hepatocellular carcinoma
* other causes of liver disease or mixed causes (excessive alcohol consumption,
* autoimmune liver disease
* immunosuppressive drugs
* infection with hepatitis C virus.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2011-08-01 (Actual); Primary Completion 2015-10-01 (Actual); Study Completion 2015-10-01 (Actual)

PRIMARY OUTCOMES:
production of protective HBsAb | three months after the last dose of vaccine
  Current treatment by NAs may suppress HBV replication but cannot completely eradicate the virus due to the systemic immune tolerance or exhaustion. HBV vaccine may enhance the immunity against HBsAg and may be an efficient immunotherapy in chronic HBV.

SECONDARY OUTCOMES:
impact on Insulin resistance, fibrosis regression | 3 month after the last dose of vaccination
  study of the possibility of improving insulin resistance and degree of fibrosis

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shaaban Hanafy A. Impact of hepatitis B vaccination on HBsAg kinetics, interferon-inducible protein 10 level and recurrence of viremia. Cytokine. 2017 Nov;99:99-105. doi: 10.1016/j.cyto.2017.08.002. Epub 2017 Aug 10. PMID 28802168